CLINICAL TRIAL: NCT01537068
Title: Desvenlafaxine (Pristiq) vs. Placebo in the Treatment of Chronic Depression
Brief Title: Desvenlafaxine vs. Placebo Treatment of Chronic Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #6457 Pfizer-WS1895577
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Dysthymic Disorder; Dysthymia; Chronic Depressive Disorder
Keywords: Dysthymic disorder; Dysthymia; Chronic non-major depression; Non-major chronic depression; Chronic depressive disorder; Antidepressant treatment
MeSH Terms: conditions — Dysthymic Disorder | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desvenlafaxine (Experimental): Serotonin-norepinephrine reuptake inhibitors (SNRIs) antidepressant drug
  Interventions: Drug: Desvenlafaxine
- Placebo (Placebo Comparator): Placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desvenlafaxine — Desvenlafaxine oral dose ranging from 50 to 100 mg/day
  Other Names: Pristiq
  Arms: Desvenlafaxine
Drug: Placebo — Matching placebo pills
  Other Names: Inactive comparator
  Arms: Placebo

SUMMARY:
The investigators are studying a new antidepressant medicine, desvenlafaxine, for the treatment of people with chronic depression. Desvenlafaxine (trade name Pristiq) has been approved by the FDA for the treatment of major depression.

The investigators are testing whether this medicine is also effective for adults with a type of chronic depression that is less severe than major depression. This condition is also known as dysthymic disorder or dysthymia. Chronic depression, lasting two or more years, often causes significant suffering and impairment.

In addition, the investigators are using MRI imaging, which uses magnetic signals to make pictures of the brain's structure and also of its functioning. The purpose of MRI imaging in this study is to see whether chronic depression is associated with differences in brain structure or functioning, and whether such differences change after medication or placebo treatment. To test this MRI scans are done at the start of the study and after 12 weeks of medication or placebo treatment. Getting MRI imaging will be an option for participants in this study but is not required.

This study involves a 6 to 12 week double-blind period during which half of the participants will take the new medication and half will take a placebo (an inactive look-alike pill). After the double blind phase, all subjects can be treated for 12 weeks with an FDA-approved antidepressant medication.

Assessments (of depressive symptoms, social functioning, and personality) will be done by study staff and by patients before the study starts, at each study visit for the first 12 weeks, and again after 24 weeks in the study.

DETAILED DESCRIPTION:
The investigators wish to study acute efficacy for 12 weeks on a double blind basis and continued response after open-label treatment at week 24 follow-up. It is important to establish the acute (12 week) efficacy of desvenlafaxine in non-major chronic depression. Also, given that non-major chronic depression is by definition chronic, it is important to demonstrate that benefit persists at follow-up assessment (24 weeks); this is clinically important in trying to alleviate the significant psychosocial morbidity associated with this disorder.

The investigators believe this study will have significant value in the treatment of patients with non-major chronic depression, and will add significantly to what remains an extremely small scientific literature.

The investigators would also like to study the effects of desvenlafaxine on brain structure and function. Learning that a medication reduces symptoms does not teach us how the medication achieves this outcome. Participants in this study can have the opportunity to participate in MRI scanning that will help to understand the mechanisms by with desvenlafaxine is effective. MRI scans are done prior to starting the clinical trial and then again after completing the double blind clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 20 to 65 years of age, inclusive
* Principal DSM-5 diagnosis of unipolar non-major Chronic Depressive Disorder (including Major Depression in partial remission, Major Depression, residual, Dysthymic Disorder, or Depressive Disorder NOS)
* Minimum of 2 years duration of the current episode of depressive disorder.
* Score of 12 or higher on the Hamilton Depression Scale (24 items) at baseline

Exclusion Criteria:

* Full remission of depression in past 24 months
* Current major depression diagnosis, psychotic illness
* Current risk of suicide
* Drug or alcohol abuse/dependence in past 6 months
* Active medical illness
* Prior nonresponse to desvenlafaxine
* Medical illness contraindicating use of desvenlafaxine
* Current or planned pregnancy during study period

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Hellerstein, MD, Principal Investigator — New York State Psychiatric Institute, Columbia University Department of Psychiatry
Locations (2):
- United States (2):
  - New York State Psychiatric Institute/3 Columbus Circle Midtown, New York, New York
  - Depression Evaluation Service (DES), New York State Psychiatric Institute, Columbia University Department of Psychiatry, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeMartinis NA, Yeung PP, Entsuah R, Manley AL. A double-blind, placebo-controlled study of the efficacy and safety of desvenlafaxine succinate in the treatment of major depressive disorder. J Clin Psychiatry. 2007 May;68(5):677-88. doi: 10.4088/jcp.v68n0504. PMID 17503976
- [Background] Levkovitz Y, Tedeschini E, Papakostas GI. Efficacy of antidepressants for dysthymia: a meta-analysis of placebo-controlled randomized trials. J Clin Psychiatry. 2011 Apr;72(4):509-14. doi: 10.4088/JCP.09m05949blu. PMID 21527126
- [Derived] Bansal R, Hellerstein DJ, Sawardekar S, Chen Y, Peterson BS. A randomized controlled trial of desvenlafaxine-induced structural brain changes in the treatment of persistent depressive disorder. Psychiatry Res Neuroimaging. 2023 Jun;331:111634. doi: 10.1016/j.pscychresns.2023.111634. Epub 2023 Mar 24. PMID 36996664
- [Derived] Yang J, Hellerstein DJ, Chen Y, McGrath PJ, Stewart JW, Peterson BS, Wang Z. Serotonin-norepinephrine reuptake inhibitor antidepressant effects on regional connectivity of the thalamus in persistent depressive disorder: evidence from two randomized, double-blind, placebo-controlled clinical trials. Brain Commun. 2022 Apr 15;4(3):fcac100. doi: 10.1093/braincomms/fcac100. eCollection 2022. PMID 35592490
- [Derived] Hellerstein DJ, Stewart JW, Chen Y, Arunagiri V, Peterson BS, McGrath PJ. Desvenlafaxine vs. placebo in the treatment of persistent depressive disorder. J Affect Disord. 2019 Feb 15;245:403-411. doi: 10.1016/j.jad.2018.11.065. Epub 2018 Nov 5. PMID 30423468
- See also: Depression Evaluation Service, NY State Psychiatric Institute website — http://www.depression-nyc.org
- See also: Columbia Psychiatry website, clinical trials — http://sklad.cumc.columbia.edu/psychiatry/clinical_trials/View_Trial.php?ID=366&type=simple

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Desvenlafaxine | Placebo
Started | 30 | 29
Completed | 26 | 26
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Population: 59 met inclusion criteria and started with study medication.
Groups:
- Desvenlafaxine: SNRI antidepressant drug
  Desvenlafaxine: Desvenlafaxine oral dose ranging from 50 to 100 mg/day
- Total: Total of all reporting groups
Arm/Group | Desvenlafaxine | Placebo | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 29 | 59
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.80 (14.18) | 36.28 (11.65) | 38.07 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 11 | 15 | 26
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression (HDRS24)
Description: HDRS-24 total score, standardly used rating scale for depression. Score 0-7 no depression; Score 8-16 mild depression; Score 17-23 moderate depression; Score 24 and up severe depression. Range= 0 to 75, higher score=worse depression
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desvenlafaxine | Placebo
Number analyzed (Participants) | 30 | 29
units on a scale | 14.63 (3.39) | 14.21 (3.50)
Statistical Analysis 1: Comparison: Desvenlafaxine vs Placebo; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis; Repeated Measures of ANOVA; Test of Within-subjects effects = 2.95

2. Primary Outcome: Hamilton Rating Scale for Depression (HDRS24)
Description: as for outcome 1
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desvenlafaxine | Placebo
Number analyzed (Participants) | 30 | 29
units on a scale | 6.53 (3.98) | 8.24 (4.86)

3. Secondary Outcome: Response Rate
Description: Assessment of overall improvement: based on HDRS and Clinical Global Improvement Scale Response Rate is defined as 50% improvement of Hamd24 summary scores from baseline.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Desvenlafaxine | Placebo
Number analyzed (Participants) | 26 | 26
Participants | 16 | 7
Statistical Analysis 1: Comparison: Desvenlafaxine vs Placebo; Test type: Superiority or Other; p = 0.025, Chi-squared; Chi-squared = 6.32

ADVERSE EVENTS:
Arm/Group | Desvenlafaxine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/29
Other Adverse Events (participants affected / at risk) | 29/30 | 19/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desvenlafaxine (N=30) | Placebo (N=29)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) — Patient was treated with placebo and this was an pre-existing condition.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desvenlafaxine (N=30) | Placebo (N=29)
Decreased sleep (Metabolism and nutrition disorders) | 10 (10) | 4 (4)
Daytime Sleepiness (Metabolism and nutrition disorders) | 9 (9) | 5 (5)
Headache (General disorders) | 9 (9) | 4 (4)
Nausea (General disorders) | 9 (9) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 7 (7) | 2 (2)
Agitation (General disorders) | 5 (5) | 0 (0)
Dizziness (General disorders) | 5 (5) | 0 (0)
Sweating (General disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No